CLINICAL TRIAL: NCT02465177
Title: Tailoring Screening, Brief Intervention, and Referral to Treatment for Medical Intensive Care Unit Survivors
Brief Title: Tailoring Screening, Brief Intervention, and Referral to Treatment for Medical ICU Survivors
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Other Study IDs: 13-3159; UL1TR001082 (NIH)
Record Dates: First submitted 2015-05-26; First posted 2015-06-08 (Estimated); Last update posted 2021-02-18 (Actual); Status verified 2021-02

CONDITIONS: Unhealthy Alcohol Use; Alcohol Use Disorders
Keywords: Unhealthy alcohol use; ICU survivors; Alcohol use disorder; SBIRT; Screening, brief intervention, and referral to treatment
MeSH Terms: conditions — Alcoholism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Unhealthy alcohol use is present in up to 38% of the 4 million patients admitted to an American intensive care unit (ICU) each year in the US. Despite the high prevalence of unhealthy alcohol use in ICU survivors, routine interventions targeted at reducing alcohol consumption, alcohol-related consequences, and illness related to alcohol are not currently part of the multidisciplinary approach to critical care. Although screening, brief intervention, and referral to treatment (SBIRT) has been described in several healthcare settings, it fails to address common characteristics of medical ICU survivors including high rates of alcohol use disorders, cognitive dysfunction, psychiatric comorbidities, and intimate involvement of friends and family. This study uses a qualitative approach to further understand the needs of medical ICU survivors with unhealthy alcohol use. The investigators hypothesize that there are common, modifiable barriers to improving alcohol-related outcomes

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older
* admitted to the medical ICU
* resolution of critical illness
* resolution of delirium/agitation
* AUDIT score 8 or greater for men, 5 or greater for women

Exclusion Criteria:

* unable to provide informed consent
* prisoner
* Unable to speak or write in English
* Pregnant

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients admitted to one of 3 medical intensive care units in the Denver metropolitan area
Sampling Method: Non-Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2014-07; Primary Completion 2021-11 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change in alcohol use | 3 months
  Change in alcohol use as assessed using a Semi-structured qualitative interview

CONTACTS AND LOCATIONS:
Locations (1):
- University of Colorado Hospital, Aurora, Colorado, United States